CLINICAL TRIAL: NCT04516616
Title: Study of Pd-1 Antibody in Combination with Neoadjuvant Chemotherapy for Locally Advanced Cervical Cancer
Brief Title: Pd-1 Antibody Combined Neoadjuvant Chemotherapy for Locally Advanced Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other); Qilu Hospital of Shandong University (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Army Medical University, China (Other); Peking University People's Hospital (Other); Tianjin Medical University General Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Chongqing University Cancer Hospital (Other); The First Affiliated Hospital of China University of Science and Technology (Anhui Provincial) (Other)
Responsible Party: Principal Investigator, Ding Ma, Director of Obstetrics and Gynecology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-S112; NACI-CERV-001 (Other: Tongji Hospital, Tongji Medical College, HUST); MA-CervC-II-002 (Other: Jiangsu Hengrui Pharmaceuticals Co., Ltd.)
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-10

CONDITIONS: Uterine Cervical Neoplasm; Uterine Cervical Cancer; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): Patients receive 1 cycle of cisplatin and albumin-bound paclitaxel combined neoadjuvant chemotherapy and subsequent 2 cycles of PD-1 antibody combined neoadjuvant chemotherapy.
  Interventions: Drug: Cisplatin+Albumin-bound paclitaxel (1 cycle) and PD-1 monoclonal antibody+Cisplatin+Albumin-bound paclitaxel (2 cycles)

INTERVENTIONS:
Drug: Cisplatin+Albumin-bound paclitaxel (1 cycle) and PD-1 monoclonal antibody+Cisplatin+Albumin-bound paclitaxel (2 cycles) — PD-1 monoclonal antibody （SHR-1210)：200mg，IV infusion，Q3W Cisplatin：75-80 mg/m2, IV infusion, Q3W Albumin-bound paclitaxel: 260 mg/m2，30min，IV infusion, Q3W

SUMMARY:
Cervical cancer is one of the major health problems for chinese women. Besides surgery and radiotherapy, neoadjuvant chemotherapy has been proved to be an effective program by many studies. However, not all patients respond well to neoadjuvant chemotherapy. This is an open-label, single-arm, multi-center clinical trial to evaluate whether PD-1 in combination with neoadjuvant chemotherapy will achieve better objective response rate.

DETAILED DESCRIPTION:
Subjects will receive therapy Q3W until evaluation of efficacy. The first cycle include cisplatin and albumin-bound paclitaxel. A combination of anti-PD-1 antibody (SHR-1210) with cisplatin and albumin-bound paclitaxel would be given in second and third cycles. Patients who have demonstrated complete or partial tumour responses （CR/PR）will receive surgery and receive postoperative adjuvant therapy in accordance with NCCN guideline. Patients who have demonstrated stable disease or progressive disease （SD/PD）will receive concurrent radiochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced (2018 FIGO staged IB3, IIA2 and IIB/IIIC1r（tumor size ≥ 4cm) ) cervical cancer and had not received any treatment before.
2. Histologically confirmed squamous carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix.
3. Pathological examination of the PD-L1 positive（Combined score Positive Score≥1）.
4. Females 18-70 years of age.
5. Eastern Cooperative Oncology Group score 0-1.
6. WBC≥3.5*10^9/L, NEU≥1.5*10^9/L, Platelet≥80×10^9 /L; AST and ALT ≤1.5 times normal upper limit; Total bilirubin ≤1.5 times the upper limit of normal value; serum creatinine and blood urea nitrogen ≤the upper limit of normal value.
7. Well-compliance and willing to keep in touch.
8. Willing to participate in this study, and sign the informed consent.

Exclusion Criteria:

1. Active or known or suspected autoimmune disease requires a system treatment as follows but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, thyroid dysfunction, asthma requiring intervention with bronchodilators.
2. HIV infection, active HBV/HCV.
3. Condition requiring systemic treatment with small doses of corticosteroids within 1 months or large doses of corticosteroids within 3 months prior to randomization.
4. Any primary malignancy within 5 years.
5. Participate in other drug clinical trials at the same time.
6. Pregnant or lactating female patients.
7. Comorbidity including but not limited to: heart diseases (grade III-IV cardiac insufficiency (NYHA standard); central nervous system diseases or nonfunctional behavior; hematological system diseases; liver or kidney malformation or history of surgery.
8. Drug or alcohol abuse.
9. Unable or unwilling to sign informed consents.
10. Not eligible for the study judged by researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 3 months
  ORR is defined as the percentage of the participants in the ITT population who have a Complete Response or Partial Response. The ORR will be assessed by a blind independent central reviewer per RECIST 1.1

SECONDARY OUTCOMES:
Pathological response rate | 3 months
  Pathological response rate is defined as the percentage of the participants in the ITT population who have complete pathologic remission or the infiltration depth of cervical lesions was < 3mm in histological examination.
Event-free survival (EFS) | 5 years
  EFS defined as the time interval from the date of participation to disease progression, local or distant recurrence (in patients undergoing surgery), or death due to any cause.
Overall survival （OS） | 5 years
  OS is defined as the time from the date of participation until death.

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, M.D., PhD, Study Chair — Tongji Hospital, Tongji Medical College, HUST
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years after completion of the study
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.

REFERENCES:
- [Derived] Li K, Chen J, Hu Y, Wang YZ, Shen Y, Chen G, Peng W, Fang Z, Xia B, Chen X, Song K, Wang Y, Zou D, Wang YC, Han Y, Feng X, Yuan J, Guo S, Meng X, Feng C, Chen Y, Yang J, Fan J, Wang J, Ai J, Ma D, Sun C. Neoadjuvant chemotherapy plus camrelizumab for locally advanced cervical cancer (NACI study): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2024 Jan;25(1):76-85. doi: 10.1016/S1470-2045(23)00531-4. Epub 2023 Dec 1. PMID 38048802
- [Derived] Fan J, Lu F, Qin T, Peng W, Zhuang X, Li Y, Hou X, Fang Z, Yang Y, Guo E, Yang B, Li X, Fu Y, Kang X, Wu Z, Han L, Mills GB, Ma X, Li K, Wu P, Ma D, Chen G, Sun C. Multiomic analysis of cervical squamous cell carcinoma identifies cellular ecosystems with biological and clinical relevance. Nat Genet. 2023 Dec;55(12):2175-2188. doi: 10.1038/s41588-023-01570-0. Epub 2023 Nov 20. PMID 37985817
- [Derived] Chen J, Han Y, Hu Y, Feng X, Meng X, Guo S, Sun C, Chen G, Li K. Neoadjuvant camrelizumab plus chemotherapy for locally advanced cervical cancer (NACI Study): a study protocol of a prospective, single-arm, phase II trial. BMJ Open. 2023 May 30;13(5):e067767. doi: 10.1136/bmjopen-2022-067767. PMID 37253491